CLINICAL TRIAL: NCT00851474
Title: Measurement of Cardiac Output and Blood Volumes
Acronym: WSU
Status: Withdrawn | Type: Observational
Why Stopped: Protocol not renewed
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-COSTATUS-7A-H; 2R44HL061994-04A2 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output
Keywords: COstatus(R); Ultrasound Dilution; Cardiac Output; Blood Volumes; Comparison of COstatus(R) cardiac output with other methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac Output (amount of blood pumped by the heart in one minute) will be measured using the new COstatus(R) system and these values will be compared with cardiac output values measured by other methods such as thermodilution. Blood volumes measured by the COstatus(R) system will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years of age)
* Should have both arterial and central venous catheters already in place

Exclusion Criteria:

* Patients who do not have either the arterial or central venous catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (older than 18 years of age) in the Intensive Care Unit with arterial and central venous catheters in place.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Compare cardiac output measured by COstatus(R) with other methods such as PA Thermodilution | 5-8 minutes minimum

SECONDARY OUTCOMES:
Measure blood volumes | 5-8 minutes minimum

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Diebel, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416